CLINICAL TRIAL: NCT00952523
Title: An Investigator-Blind, Phase 4 Study Assessing the Facial Irritation Potential of Two Acne Treatment Products (Retin-A Micro Gel, 0.04% Pump and Epiduo Gel) Using a Split-Face Model
Brief Title: Evaluation of Irritation That Potentially Could be Caused by Two Facial Gels Applied to Opposite Sides of the Face
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CA-P-7190
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2010-04-09 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Acne Vulgaris
Keywords: acne; irritation; objective sensory methods
MeSH Terms: conditions — Acne Vulgaris | interventions — Tretinoin; Adapalene

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tretinoin & Adapalene-Benzoyl Peroxide (Experimental): Tretinoin and Adapalene-Benzoyl Peroxide facial gels applied once daily in a split face model
  Interventions: Drug: Tretinoin Facial Gel; Drug: Adapalene/Benzoyl Peroxide Facial Gel

INTERVENTIONS:
Drug: Tretinoin Facial Gel — A marketed facial gel containing Tretinoin 0.04% is applied to one side of the face daily for three weeks.
  Other Names: Retin-A Micro Gel 0.04% Pump
Drug: Adapalene/Benzoyl Peroxide Facial Gel — A marketed facial gel containing Adapalene .1% and Benzoyl peroxide 2.5% is applied to the other side of the face daily for three weeks
  Other Names: Epiduo Gel

SUMMARY:
A study to compare the skin irritation potential of two marketed gels for acne treatment, each applied to half of the face of healthy volunteers.

DETAILED DESCRIPTION:
At the Baseline Visit, following satisfaction of entry criteria and screening procedures, all subjects will be applying two products to their faces, each on one side only. The side of the face receiving each product is randomly assigned. One group will use Retin-A MICRO Gel, (tretinoin) 0.04% Pump on the left side of the face and Epiduo Gel (adapalene .1% and benzoyl peroxide 2.5%), on the right side of the face daily for 3 consecutive weeks after washing with study-supplied facial wash. The other group will use the same products, but on opposite sides of the face for three consecutive weeks after washing with the same study-supplied facial wash.

Subjects will return to the study center every weekday morning for evaluation and application of both study products. Applications done on the weekends, will be done at home by the subject. At each visit the subject will be scored for cutaneous treatment effects by a blinded evaluator. At baseline and at the end of each week, subjects will be photographed and have chromometer readings.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Before screening, subjects (or legally authorized representative) must read and sign the IRB approved Informed Consent Form (includes HIPPA and Photo release)
* Subjects must have Fitzpatrick Skin Type I, II or III, and judged by the Investigator to have healthy skin
* Subject's bilateral facial skin must be clear of any confounding irritation, rashes, acne, rosacea, etc. prior to the study
* Subject must be free of systemic retinoids for at least 2 months
* Subject must not be using any topical retinoids, systemic antibiotics, nicotinamide or systemic steroids for 1 month prior to study start
* All other topical medications to face (e.g., steroids, antimicrobials, salicylic acid and benzoyl peroxide) and cosmetics containing retinols, AHA's and bleaching agents such as hydroquinone are to be discontinued at least 2 weeks prior to study initiation
* Subjects will not apply any emollients and cosmetics to the facial area 24 hours prior to study initiation
* Subject must not be planning to become pregnant or nursing before entering the study and during the study period. In addition if using birth control pills, subject must be stabilized for at least 2 months. If subject is of child bearing potential, subject must be using approved method of birth control. Approved methods are birth control pills, implants, patches or spermicide with condoms.

Exclusion Criteria:

* Subjects who are pregnant or nursing
* Subjects who have a grade 1 or more for facial erythema
* Subjects who exhibit any skin condition (i.e., atopic dermatitis, seborrheic dermatitis, and psoriasis) or disease that may require concurrent therapy or may confound the evaluation of drug safety or efficacy
* Subjects who have a history of hypersensitivity to any of the formulation components
* Subjects who have received any experimental drug or used any experimental device 30 days prior to initiation of study therapy
* Subjects who have excessive facial hair that may obstruct or hinder the evaluation of any reactions
* Subjects who use any known photosensitizing agents
* Subjects who presently have skin cancer or actinic keratosis on the face

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Lineberry, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Skin Study Center, Broomall, Pennsylvania, United States

REFERENCES:
- [Result] Leyden JJ, Nighland M, Rossi AB, Ramaswamy R. Irritation potential of tretinoin gel microsphere pump versus adapalene plus benzoyl peroxide gel. J Drugs Dermatol. 2010 Aug;9(8):998-1003. PMID 20684151
- See also: FDA's Drug Finder — http://www.accessdata.fda.gov/scripts/cder/drugsatfda/index.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tretinoin & Adapalene-Benzoyl Peroxide
Started | 162
Completed | 155
Not Completed | 7
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Arm/Group | Tretinoin & Adapalene-Benzoyl Peroxide
Number analyzed (Participants) | 162
Age Continuous [Mean (Standard Deviation); unit: years] | 31 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 162

OUTCOME MEASURES:

1. Primary Outcome: Facial Irritation and Cutaneous Effects
Description: Scores on a scale were recorded each weekday. The scale for Erythema and Dryness was from 0=none to 8=severe (highest possible score is calculated as 8x5daysx3weeks=120). The scale for Burning/Stinging and Itching was from 0=none to 3=severe (highest possible score was calculated as 3x5daysx3weeks=45). The scores that were accumulated through the study for each treatment were then compared.
Time Frame: three weeks
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Groups:
- Tretinoin Facial Gel: Tretinoin facial gel in a 0.04% Pump
- Adapalene-Benzoyl Peroxide Facial Gel: Adapalene 0.1% and Benzoyl peroxide 2.5%
Arm/Group | Tretinoin Facial Gel | Adapalene-Benzoyl Peroxide Facial Gel
Number analyzed (Participants) | 162 | 162
Scores on a Scale
  Erythema | 1.5 (3.8) | 5.4 (11.8)
  Dryness | 3.1 (6.1) | 7.8 (10.3)
  Burning/Stinging | 1.9 (4.0) | 5.8 (6.5)
  Itching | 1.0 (2.3) | 2.9 (4.4)

ADVERSE EVENTS:
Groups:
- Tretinoin Facial Gel: Tretinoin facial gel applied once daily in a split face model
- Adapalene-Benzoyl Peroxide Facial Gel: Adapalene-Benzoyl Peroxide facial gel applied once daily in a split face model
Arm/Group | Tretinoin Facial Gel | Adapalene-Benzoyl Peroxide Facial Gel
Serious Adverse Events (participants affected / at risk) | 0/162 | 0/162
Other Adverse Events (participants affected / at risk) | 0/162 | 0/162

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less